CLINICAL TRIAL: NCT07000604
Title: Effect of Inhaler Medication Use on Oral Health in COPD Patients: A Randomized Controlled Trial
Brief Title: Effect of ınhaler Use on Oral Health in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Betül YALÇIN, NURSE, Çankırı Karatekin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-07-2024-15-COPD01
Record Dates: First submitted 2025-05-15; First posted 2025-06-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: EXPERIMENTAL AND CONTROL GROUP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DENEY GRUBU (Other): Oral care training will be given to 40 randomly selected patients and their oral health will then be evaluated.
  Interventions: Other: Mouth Care Training

INTERVENTIONS:
Other: Mouth Care Training — Patients will be educated on how to care for their mouths after using inhaled medication.

SUMMARY:
The aim of this study was to evaluate the effect of oral health education given to individuals diagnosed with COPD and using inhaled medication.

DETAILED DESCRIPTION:
Before the research data are collected, the purpose, content, scope and duration of the research will be explained in one-to-one interviews with the participants. Verbal and written informed consent will be obtained from the participants. After the participants gave consent to the study, they will be divided into intervention and control groups by simple random sampling method. Participants will be asked to answer the questions in the data collection tools as they see fit and to answer all of the questions. The data collection form will be applied through face-to-face interviews with participants who meet the inclusion criteria. After each completed questionnaire, the researchers will check whether the answers to the survey questions are missing. When unanswered questions are identified, participants will be invited to fill in the missing information. The completion of the questionnaires and training is planned to take an average of 20-25 minutes for each participant. The experimental group will receive training intervention. No education will be given to the control group. After 3 months, an appointment will be made to evaluate oral health

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD for at least 6 months,
* Outpatient and inpatient,
* Consent to participate in the research,
* Not under the age of eighteen,
* With a metered dose inhaler (MDI) in treatment,
* No communication barriers,
* No COPD exacerbation and/or respiratory tract infection,
* According to the GOLD report; mild (Stage 1), moderate (Stage 2), severe (Stage 3).

Exclusion Criteria:

* Diagnosed with COPD for less than 6 months,
* Refused to participate in the research,
* Treatment without metered dose inhalers (MDIs),
* Uncommunicative,
* Those who withdrew from participating in the study during data collection,
* Not completing the survey,
* COPD exacerbation and/or respiratory tract infection,

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Oral Health Status with Oral Assessment Guide | Baseline and 3 months after intervention
  Oral health status will be assessed using the Oral Assessment Guide. After the training, the scores of the trained group and the untrained group will be compared to determine the effect of oral care training. Each change in oral health is scored between 1 and 3 points and these points are added to obtain a total score. The guide supports the creation of an oral care protocol for a patient with a deteriorated oral mucous membrane. The scores that can be obtained from the guide vary between 8 and 24. A total oral mucous membrane score (OMP) between 8 and 14 indicates "oral-mucous membrane deterioration risk", while a score between 14 and 24 indicates "oral mucous membrane deterioration". According to the oral assessment guide, individuals with low scores indicate that their oral health is good, while high scores indicate a negative change in oral health.

SECONDARY OUTCOMES:
Medication Adherence with Medication Adherence Reporting Scale | Baseline and 3 months after intervention
  Patients' compliance with inhaler use will be assessed using the Medication Adherence Reporting Scale. There are 5 items in the scale. A 5-point Likert-type scale (1=always, 5=never) is used for responses. The scores that can be obtained from the scale vary between 5 and 25. An increase in the total score of the scale indicates increased medication compliance, while a decrease in the score indicates decreased medication compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yalçın, 2, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Çankiri Devlet Hastanesi, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No